CLINICAL TRIAL: NCT01770301
Title: A Randomized, Open Label, Phase II Trial of Bevacizumab Plus Weekly Paclitaxel Followed by Bevacizumab Monotherapy Maintenance Versus Weekly Paclitaxel Followed by Observation in Patients With Relapsed Ovarian Sex-cord Stromal Tumours
Brief Title: Efficacy and Safety of Bevacizumab (Avastin®) Combined to Weekly Paclitaxel Followed by Bevacizumab (Avastin®) Alone in Patients With Relapsed Ovarian Sex-cord Stromal Tumours (ALIENOR)
Acronym: ALIENOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALIENOR (GINECO-OV222)
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Ovarian Sex-cord Stromal Tumor
MeSH Terms: interventions — Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A - Paclitaxel (Active Comparator): patients will receive paclitaxel alone at the dose 80 mg/m² administered by intravenous injection at D1, D8 and D15 every 4 weeks for 6 cycles. Thereafter, patients will be followed-up with imaging exams every 12 weeks. At the time of confirmed progression, patients could receive bevacizumab 15 mg/kg every 3 weeks for 12 months following investigator's decision. In some cases, longer therapy may be allowed after discussion with the Principal Investigator/Sponsor
  Interventions: Drug: Paclitaxel
- B - Paclitaxel + Bevacizumab followed by Bevacizumab (Experimental): patients will receive paclitaxel at the dose 80 mg/m² administered by intravenous injection at D1, D8 and D15 every 4 weeks + Bevacizumab at the dose 10 mg/kg administered by intravenous injection every 2 weeks (D1 and D15) for 6 cycles. Thereafter, patients will receive IV injection of bevacizumab 15 mg/kg every 3 weeks for up to 1 year
  Interventions: Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Paclitaxel
Drug: Bevacizumab
  Arms: B - Paclitaxel + Bevacizumab followed by Bevacizumab

SUMMARY:
Bevacizumab (called also Avastin ®) is a medicine preventing the creation of new blood vessels (a process called "angiogenesis"). This can reduce blood flow of the tumor and then decreasing the contribution of nutriments and oxygen to the cancer cells and prevent the tumor from growing.

In various types of cancers, as lung, breast, colorectal and renal cancer, addition of the bevacizumab to chemotherapy allowed to improve the disease outcome. The bevacizumab already benefits from a marketing authorization (MMA) for these various types of cancers.

The bevacizumab has also obtained MMA for the treatment of the ovarian cancer in its most frequent histological form (ovarian carcinoma). Clinical trials conducted in this indication demonstrated the importance to pursue the treatment by bevacizumab after the chemotherapy is ended.

This anti-angiogenic medicine is thought to be of a potential interest in sex cords- stromal since this tumors are very well vascularized.

The ALIENOR study aims to explore the interest and the clinical benefit of associating bevacizumab to the paclitaxel in order to treat patients suffering from recurring sex cords- stromal tumor treated beforehand by platinum chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥ 18 years at inclusion
* Histologically confirmed diagnosis of ovarian Sex cord-stromal tumors including the following cell types: granulosa cell tumours (adults and juveniles types), granulosa cell-theca cell tumour, Sertoli-Leydig cell tumours, malignant steroid cell tumours, gynandroblastoma, unclassified SCST and mixed tumours
* Documented relapse of SCST defined by progression of disease (radiologic, clinic or biological progression)
* At least one measurable site of disease as defined by RECIST 1.1

  * Tumours within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence > 90 days following completion of radiotherapy.
* Patients must have been pre-treated with at least 1 prior line of platinum-based chemotherapy
* Adequate bone marrow, liver and renal functions including the following:

  * Absolute neutrophil count ≥ 1.5 G/L, platelet count ≥ 100 G/L, and hemoglobin ≥ 9 g/dL. Prior transfusion is authorized to keep haemoglobin level to ≥9g/dL
  * AST/ALT ≤ 3 x upper limit of normal (ULN) (or ≤ 5.0 ULN if liver metastasis) and total bilirubin ≤ 1.5 ULN
  * Serum creatinine ≤ 1.5 ULN or calculated creatinine clearance ≥ 50 mL/min according to Cockcroft formula (or to MDRD formula for patients older than 65 years-old).
* Adequate coagulation panel:

  * PT ≤ 1.2 ULN
  * aPTT ≤ 1.5 ULN
  * INR ≤ 1.5 ULN
* Adequate neurologic function: only neuropathy (sensory and motor) grade ≤ 1 (CTCAE v4.3) are allowed
* ECOG Performance status of 0, 1, or 2 (Appendix 5)
* Life expectancy ≥ 4 months
* Satisfactory cardiac function
* Ability to understand and sign informed consent and willingness to comply with the study procedures before study entry
* Women of childbearing potential* are required to have a negative serum pregnancy test within 7 days prior to study treatment initiation (i.e. Cycle 1 Day 1) and are willing to use adequate contraceptive method during the whole study period and for up to 6 months after the last treatment intake

  *: Female patients who meet at least one of the following criteria are defined as women of non-childbearing potential:
  * ≥ 50 years old and naturally amenorrheic for ≥ 1 year
  * Permanent premature ovarian failure confirmed by a specialist gynaecologist

    * Previous bilateral salpingo-oophorectomy or hysterectomy
    * XY genotype, Turner's syndrome, or uterine agenesis
    * Female patient who do not meet at least of the above criteria are defined as women of childbearing potential
* Covered by a medical insurance (in country where applicable)

Exclusion Criteria:

* Prior systemic therapy with bevacizumab
* Active peripheral neuropathy ≥ grade 3 (NCI-CTCAE v4.3)
* Prior history of other malignancies other than ovarian SCST (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the subjects has been free of the disease for at least 3 years or 5 years for breast cancer
* No resolution of specific toxicities related to any prior anti-cancer therapy to grade ≤1, excluding alopecia, according to the NCI-CTCAE v.4.3
* History or evidence of thrombotic or hemorrhagic disorders, including cerebro-vascular accident/stroke or transient ischemic attack or sub-arachnoids' haemorrhage within 6 months prior to first dose of study drugs
* Uncontrolled arterial hypertension (systolic ≥ 150 mmHg or diastolic ≥ 100 mmHg) despite optimal antihypertensive therapy or clinically significant cardiovascular disease including one of the following:

  * Myocardial infarction or instable angina within 6 months prior to first dose of study drugs
  * NYHA grade ≥ II congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Peripheral vascular disease ≥ grade 3
* History of bowel obstruction, including sub-occlusive syndrome and history of abdominal fistula, gastro-intestinal perforation or intra-abdominal abscess during the year prior to inclusion
* Prior treatments:

  * Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study inclusion or anticipation of need for major surgical procedure during the course of the study
  * Current or recent treatment with another investigational drug within 30 days of first study treatment dosing or within 6 weeks in case of prior nitrozo-urea and or mitomycin C treatment. In case of hormonotherapy , patients will be eligible if hormonotherapy is discontinued within at least 1 week before treatment initiation
  * Current or recent (within 10 days prior to randomization) chronic use of aspirin> 325 mg/day or use of any other inhibitor of platelet aggregation
  * Chronic treatment (i.e. > 15 days) with non steroids anti-inflammatory agents unless a washout period of 15 days was observed before the inclusion.
  * Intake of granulocyte growth factor within 3 weeks before study entry
* Presence of hematuria and proteinuria ≥ 2+ (urine dipstick). Patients with ≥ 2+ proteinuria on dipstick at screening should undergo a 24-hour urine collection and will be eligible only if 24-h proteinuria ≤ 1 g
* Untreated evolutive brain metastases
* Active bacteria or fungal infection (grade ≥2, CTC AE V4.3)
* Known HIV1, HIV2 or chronic hepatitis B or C infection
* Hypersensitivity to Chinese hamster ovary (CHO) cell products or other recombinant human or humanized antibodies
* Any contraindications to paclitaxel treatment: for example severe hypersensitivity reactions to paclitaxel, macrogolglycerol ricinoleate (polyoxyl castor oil) or to any of the excipients (Ethanol Citric acid) (refer to Taxol® SPC for further details)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
clinical benefit of combining bevacizumab treatment to weekly paclitaxel | after 6 months of treatment
  To evaluate the clinical benefit of combining bevacizumab treatment to weekly paclitaxel measured by the non-progression rate after 6 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle RAY-COQUARD, MD, PhD, Principal Investigator — Centre Léon Bérard, LYON, FRANCE
Locations (24):
- France (24):
  - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - ICM Val d'Aurelle, Montpellier
  - ORACLE - Centre d'Oncologie de Gentilly, Nancy
  - Hôpital Privé du Confluent, Nantes
  - Hôpital Cochin, Paris
  - Groupe Hospitalier Diaconesses - Croix Saint-Simon, Paris
  - Hôpital Tenon, Paris
  - Centre CARIO - HPCA, Plérin
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - ICO Centre René Gauducheau, Saint-Herblain
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - ICL Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Ray-Coquard I, Harter P, Lorusso D, Dalban C, Vergote I, Fujiwara K, Gladieff L, Luck HJ, Floquet A, Chevalier-Place A, Schnelzer A, Pignata S, Selle F, Sehouli J, Brocard F, Mangili G, Pautier P, De Giorgi U, Provansal M, Heudel PE. Effect of Weekly Paclitaxel With or Without Bevacizumab on Progression-Free Rate Among Patients With Relapsed Ovarian Sex Cord-Stromal Tumors: The ALIENOR/ENGOT-ov7 Randomized Clinical Trial. JAMA Oncol. 2020 Dec 1;6(12):1923-1930. doi: 10.1001/jamaoncol.2020.4574. PMID 33030515